CLINICAL TRIAL: NCT00165230
Title: A Phase II Study of Thalidomide in Combination With Temodar in Patients With Metastatic Neuroendocrine Tumors
Brief Title: Thalidomide in Combination With Temodar in Patients With Neuroendocrine Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other); Beth Israel Deaconess Medical Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02-011
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2009-04-28 (Estimated); Status verified 2009-04

CONDITIONS: Neuroendocrine Tumor
Keywords: thalidomide; temodar; metastatic neuroendocrine tumor; unresectable neuroendocrine tumor
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Thalidomide; Temozolomide

INTERVENTIONS:
Drug: Thalidomide
Drug: Temodar

SUMMARY:
The purpose of this study is to find out what effects, good or bad, that thalidomide and temodar have on patients with neuroendocrine tumors.

DETAILED DESCRIPTION:
* Patients will receive thalidomide orally once daily continuously unless they experience significant side effects. Temodar is given orally once a day for one week, followed by a one week break period. This one week on/one week off schedule will continue for the duration of treatment unless there are significant side effects.
* After eight weeks (2 cycles) a CT scan will be performed to see how the treatment has affected the patient's tumor. Patients will continue taking the study drug unless there is evidence of tumor growth.
* Regular blood tests will be done weekly during the first two months to make sure that the treatment is not resulting in serious side effects. If there are no side effects during the first two months, the blood tests may decrease in frequency to every two weeks.
* Immediately after the patient has completed the study they will be evaluated by physical exam, blood work, and a CT scan. The follow-up will consist of clinic visits and phone calls every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed locally unresectable or metastatic neuroendocrine tumor excluding small cell carcinoma
* Prior treatment with chemoembolization or cryotherapy is allowed
* Radiotherapy is allowed if completed more than 4 weeks prior to study.
* Measurable disease as defined by RECIST criteria
* Age greater than or equal to 18 years.
* ECOG performance status of less than or equal to 2
* ANC >1,500/mm3
* Platelet Count > 100,000/mm3
* Hemoglobin > 9 g/dl
* Serum creatinine < 1.5 x ULN
* Total bilirubin < 2 x ULN
* SGOT and SGPT < 2 x ULN
* Alkaline phosphatase < 2 x ULN
* Life expectancy of greater than 12 weeks

Exclusion Criteria:

* Clinically symptomatic central nervous system metastases or carcinomatous meningitis
* Myocardial infarction in past 6 months
* Major surgery in past two weeks
* Uncontrolled serious medical or psychiatric illness
* Insufficient recovery from all active toxicities of prior therapies
* Active nonmalignant systemic disease
* Frequent vomiting or medical condition that could interfere with oral medication intake
* Known HIV positivity or AIDS-related illness
* Pregnant or nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32
Dates: Start 2002-05; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
To assess the response rate in patients with locally unresectable neuroendocrine tumors treated with temodar and thalidomide.

SECONDARY OUTCOMES:
To evaluate overall response and progression free survival of this patient population
to evaluate the safety of temodar and thalidomide.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew H. Kulke, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconness Medical Center, Boston, Massachusetts